CLINICAL TRIAL: NCT00725582
Title: The Effects of IMA-026 on Allergen-Induced Airway Responses and Airway Inflammation in Subjects With Mild Atopic Asthma
Brief Title: Study Evaluating the Effect of IMA-026 on Allergen-Induced Late Asthma Response in Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3192K1-1002
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: IMA-026
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IMA-026
  Arms: A
Other: Placebo
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the effect of IMA-026, an antibody to IL-13, on airway hyperresponsiveness and airway inflammation in mild asthmatics. IMA-026 will be given as 2 injections under the skin 1 week apart at 2 mg/kg each dose. The study will include a screening period and a treatment period which includes doses on day 1 and day 8.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women 18 to 60 yrs with mild allergic asthma
2. only asthma med is short-acting bronchodilator used not more than twice weekly
3. FEV1 greater than 70% predicted and a demonstrated baseline late response to allergen induction

Exclusion Criteria:

1. Upper respiratory infection or asthma exacerbation with 4 weeks of screening
2. Serious infection requiring parenteral antibiotics or hospitalization with 4 weeks of test article administration
3. Positive radiographic findings indicative of respiratory disease other than asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the maximum change in FEV1 from baseline for the LAR between IMA-026 and placebo | 11 weeks

SECONDARY OUTCOMES:
Treatment comparison of the hour 3 and hour 7 FEV1 AUC for the LAR; various comparisons of the methacholine PC20 | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, Cockcroft DW, Fitzgerald JM, Carlsten C, Davis BE, Deschesnes F, Duong M, Durn BL, Howie KJ, Hui L, Kasaian MT, Killian KJ, Strinich TX, Watson RM, Y N, Zhou S, Raible D, O'Byrne PM. Effects of interleukin-13 blockade on allergen-induced airway responses in mild atopic asthma. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1007-14. doi: 10.1164/rccm.201008-1210OC. Epub 2010 Nov 5. PMID 21057005